CLINICAL TRIAL: NCT07293585
Title: Vascular Optimized Radiotherapy Tuned to Critical Structures for Erectile Function Using High-Precision X-Ray Treatment
Acronym: VORTEX
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Viewray Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 25-2129
Record Dates: First submitted 2025-12-16; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer
Keywords: sexual function
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: magnetic resonance angiography (MRA) guided active aid in identifying and avoiding internal pudendal arteries, corpora cavernosa and neurovascular bundles sensitive structures during SBRT.
Who Masked: Participant
Masking Description: single blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Arm 1 non-adaptive SBRT (Active Comparator): Patients undergo MRI or CT-guided SBRT without daily plan adaptation once every other day or on consecutive days if necessary, for a total of 5 treatments over 18 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo MRI and CT during screening and blood sample collection throughout the trial.
  Interventions: Radiation: Neurovascular sparing stereotactic body radiation therapy
- Arm 2 Neurovascular sparing stereotactic body radiation therapy (Experimental): Patients undergo MRI or CT-guided SBRT with daily plan adaptation once every other day or on consecutive days if necessary, for a total of 5 treatments over 18 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo MRI and CT during screening and blood sample collection throughout the trial.
  Interventions: Radiation: Neurovascular sparing stereotactic body radiation therapy

INTERVENTIONS:
Radiation: Neurovascular sparing stereotactic body radiation therapy — Use of adaptive radiotherapy

SUMMARY:
With people living longer after being treated for prostate cancer, quality of life has become a concern when considering the treatment plan. Sometimes after radiation therapy, patients may experience problems that affect the urinary and bowel systems, along with sexual function.

Stereotactic body radiotherapy (SBRT) is a type of radiation technique that delivers five high doses of radiation. At University of California at Los Angeles (UCLA), we have the option to administer SBRT in both our CT-guided and MRI-guided radiation machines.

This trial aims to determine the most effective method for protecting the nerves and blood vessels essential for erectile function, utilizing a technique known as neurovascular sparing.

This technique uses images (i.e., MRI) to map the neurovascular bundles of nerves and blood vessels, which are crucial for erectile function. "Adapting" the radiotherapy treatment for each of these five treatment sessions could enable a more precise delivery of your radiation treatment that is customized based on your internal anatomy immediately before the treatment starts. This is also a standard and low-risk intervention used in many different types of cancer. However, it is a very labor-intensive and time-consuming procedure that requires a team of experts to work together before each of your radiotherapy sessions. We are unsure if the increased complexity associated with this adaptive treatment reduces side effects.

DETAILED DESCRIPTION:
The mechanism implicated in sexual function decline following radiotherapy involves injury to vascular structures surrounding the prostate which are critical for normal erectile function, namely the corpora cavernosa, internal pudendal arteries, and neurovascular bundles. These structures are all in close proximity to the prostate gland and are often included at least partially within the planning target volume margin of treatment plans. As noted above, these planning target volume (PTV) expansions were historically large due to the need to ensure adequate coverage of the target volume to achieve disease control although this likely came at the cost of higher rates of treatment-related toxicity. With enhanced technology for target visualization and intra-fraction motion management, it is technically feasible to reduce margins and spare surrounding normal tissue from receiving the full prescription dose while still treating the target volume with high confidence.

Beyond reducing the isometric PTV expansion due to increased precision in radiation delivery with modern techniques, however, it is now technically feasible to crop out these sensitive Organs-at-risk (OARs) from the final PTV volume in order to further spare them from receiving excess dose. This process, referred to as neurovascular-sparing (NV-sparing), involves the fusion of an MRI and/or MR angiogram to standard radiation planning images to allow accurate contouring of the internal pudendal arteries and neurovascular bundles so that these can be intentionally spared. Daily online adaptive replanning may also play a role in ensuring appropriate coverage of the target volume and sparing of OARs as intended by the treatment plan. To date, no investigations have reported on the clinical or dosimetric outcomes of patients treated with an NV approach in conjunction with these other methods. Furthermore, specific dose constraints for these structures are largely unknown due to the lack of empiric evidence to guide selection.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18.
2. Histologically confirmed, clinically localized adenocarcinoma of the prostate.
3. Staging workup as recommended by the National Comprehensive Cancer Network (NCCN) on the basis of risk grouping.

   a. Advanced imaging studies (i.e. prostate-specific membrane antigen [PSMA] positron emission tomography [PET]/CT and fluciclovine PET/CT scan) can supplant a bone scan if performed first.
4. No evidence of metastatic disease in lymph nodes above the bifurcation of the renal arteries, or in bones or visceral organs (nodal disease identified on a PSMA PET/CT scan below the bifurcation of the renal arteries is allowable).
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤2.
6. Ability to undergo magnetic resonance angiography (MRA) of the pelvis.
7. No indication for urgent or emergent radiation.
8. Written informed consent obtained from participant or participant's legal representative and ability for participant to comply with the requirements of the study.

Exclusion Criteria:

1. Patients with neuroendocrine or small cell carcinoma of the prostate.
2. Patients with any evidence of distant metastases except that evidence of lymphadenopathy below the level of the renal arteries can be deemed locoregional per the discretion of the investigator.
3. Evidence of intraprostatic lesion by biopsy, MRI, or PSMA PET/CT within the middle third, or both lateral thirds of the prostate gland.
4. History of whole-gland cryosurgery, high-intensity focused ultrasound (HIFU), brachytherapy, or other ablative treatments of the whole prostate.
5. Prior pelvic radiotherapy.
6. History of Crohn's disease, ulcerative colitis, or ataxia telangiectasia.
7. Penile prosthesis or implant present prior to treatment.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate is required to treat
Enrollment: 200 (Estimated)
Dates: Start 2025-12-16 (Actual); Primary Completion 2035-12-16 (Estimated); Study Completion 2036-12-16 (Estimated)

PRIMARY OUTCOMES:
Expanded Prostate Cancer Index Composite (EPIC-26) sexual function Questionnaire | 24 months
  The primary endpoint is clinically relevant (≥24 point) decline in EPIC-26 sexual function domain scores at 24 months following treatment in patients randomized to NV-sparing SBRT relative to patients randomized to conventional SBRT without explicit NV-sparing.

SECONDARY OUTCOMES:
Clinically relevant acute change in International Prostate Symptom Score (I-PSS) domain of EPIC-26. | From initiation to 90 days post treatment
  Clinically relevant acute changes (from initiation to within 90 days after completion of SBRT) in IPSS of EPIC-26 patient-reported QOL. The International Prostate Symptom Score (I-PSS) is based on answers to seven questions concerning urinary symptoms and one question concerning quality of life. Answers are assigned points from 0 to 5. The total score range is from 0 -35. 0 indicating no symptoms to 35 indicating extremely symptomatic.
Clinically relevant acute change in Sexual Health Inventory for Men (SHIM) domain of EPIC-26. | From initiation to 90 days post treatment
  Clinically relevant acute changes (from initiation to within 90 days after completion of SBRT) in SHIM domain of EPIC-26 patient-reported QOL. The SHIM score range is from 5 to 25. Higher score indicates better erectile function.
Clinically relevant chronic changes in IPSS, of EPIC-26. | From initiation to 90 days post treatment
  Clinically relevant chronic changes (from initiation to within 90 days after completion of SBRT) in IPSS domain of EPIC-26 patient-reported QOL
Clinically relevant chronic changes in SHIM, of EPIC-26. | From initiation to 90 days post treatment
  Clinically relevant chronic changes (from initiation to within 90 days after completion of SBRT) in SHIM domain of EPIC-26 patient-reported QOL
Gastric ulcer (GU) or Gastriointestinal (GI) toxicity | From initiation to 90 days post treatment
  Incidence of GU or GI toxicity of at least grade 2 by the physician-reported CTCAE criteria.
prostate specific antigen (PSA) completed response at 2 years | From initiation to 90 days post treatment
  PSA completed response at 2 years, defined as proportion of patients with PSA <20% of the pre-SBRT PSA.
Biochemical Recurrence-Free Survival rate | From initiation to 90 days post treatment
  Biochemical Recurrence-Free Survival rates at 5 years, where biochemical recurrence is defined as serum PSA levels 2 ng/mL higher than the post-treatment PSA nadir.

CONTACTS AND LOCATIONS:
Overall Officials: Amar Kishan, MD, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- University of California at Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No